CLINICAL TRIAL: NCT01286857
Title: A Prospective, Open, Non-controlled Proof-of-concept Investigation to Evaluate the Function of a New Silicon Cover Film and an On-top Suction Device to be Used in a NPWT System in the Treatment of Acute and Chronic Wounds
Brief Title: An Investigation to Evaluate the Function of a New Silicon Cover Film and an On-top Suction Device to be Used in a NPWT System in the Treatment of Acute and Chronic Wounds
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Molnlycke Health Care AB (Industry)
Responsible Party: Ruth Eid-Forest, MD, Dept. of Dermatology, University Hospital of Orebro, Sweden
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SIMP 01
Record Dates: First submitted 2010-10-08; First posted 2011-01-31 (Estimated); Last update posted 2011-07-18 (Estimated); Status verified 2011-07

CONDITIONS: Acute and Chronic Wounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: External Suction Interface and a Silicon Film — Evaluate the function of a new silicon cover film and an on-top suction device to be used in a NPWT system in the treatment of acute and chronic wounds.

SUMMARY:
The aim of the investigation is to evaluate the function of two new device parts to be used in a NPWT system; an on-top suction device intended to transport exudate from the wound and a silicon cover film intended to fixate the wound filler and seal tight to the skin in order to keep a moist environment.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic wounds (venous, pressure or diabetic type), and acute wounds suitable for NPWT therapy according to the investigator's judgment
2. 1cm2 ≤ wound size ≤ 200cm2
3. Male or female, 18 years and above
4. Signed Informed Consent Form
5. Subject understands the written Patient Information

Exclusion Criteria:

1. Need for frequent dressing changes, i.e.<48 hours between the changes
2. Critical ischemia (for wound healing) according to investigator's judgement
3. Malignancy in the wound and/or wound margin
4. Target ulcer previous not successfully treated with NPWT within 48 hours
5. Poorly controlled diabetes according to investigators judgement.
6. Osteomyelitis which has been left untreated
7. Infection which has been left untreated
8. High risk for bleeding complications
9. Exposed blood vessels, organs or nerves
10. Current or within 3 months treatment with chemotherapy or irradiation
11. Known hypersensitivity to the dressing material
12. Expected technically impossible to seal the film to achieve a vacuum treatment
13. Expected non compliance with the Clinical Investigation Plan (CIP)
14. Pregnancy
15. Subjects not suitable for the investigation according to the investigator's judgement
16. Subjects previously included in this investigation
17. Subjects included in other ongoing clinical investigation at present or during the past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the transport of exudate from the wound bed to canister and thus distribute negative pressure in the wound site | 144 - 288 hours

SECONDARY OUTCOMES:
To investigate the practical properties and management of the device, to evaluate the ease of use for the subject and the care giver and to assess any undesirable effects with the suction part | 144-288 hours

CONTACTS AND LOCATIONS:
Locations (3):
- Sweden (3):
  - County Hospital, Halmstad, Halmstad
  - University Hospital of Örebro, Örebro
  - Hudmottagningen, Sundsvalls sjukhus, Sundsvall